CLINICAL TRIAL: NCT05883800
Title: TNT-RECORD:Total Neoadjuvant Treatment in Rectal Cancer With On-couch Adaptive Radiotherapy
Brief Title: Total Neoadjuvant Treatment Combined With Adaptive Radiotherapy for Rectal Cancer
Acronym: TNT-RECORD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402056
Record Dates: First submitted 2023-02-24; First posted 2023-06-01 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-07

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Intervention: daily on-couch adaptive radiotherapy
  Interventions: Radiation: On-couch adaptive radiotherapy

INTERVENTIONS:
Radiation: On-couch adaptive radiotherapy — A new treatment plan, guided by volumetric images, is created at each treatment session
  Other Names: online ART

SUMMARY:
Diarrhea was the most frequently reported severe adverse event in the treatment regime of pre-operative sequential short-course radiotherapy followed by chemotherapy (so called total neo-adjuvant treatment).

This study therefore investigates the benefit of on-couch adaptation for locally advanced rectal cancer patients undergoing this treatment regime.

DETAILED DESCRIPTION:
This is a prospective single-arm study investigating the benefit of on-couch adaptation for locally advanced rectal cancer patients prescribed with pre-operative sequential short-course radiotherapy (RT) followed by Oxaliplatin-combined chemotherapy (mFOLFOX(6) or CAPOX). On-couch adaptation, where the radiation dose is tailored to the anatomy of the patient at each radiotherapy session. Firstly, the study will investigate if on-couch adaptation result in less gastro-intestinal adverse events, secondly it will reveal if this possible reduction lead to more patients being able to fulfill all cycles of prescribed chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with loco-regional advanced rectal adenocarcinoma with clinical indications for short-course with TNT chemotherapy i.e. having at least one of the following T4a, CRM+ (≤1 mm), N1c, N2 or extramural vascular invasion (EMVI+). Patients presenting at least one of these criteria in addition to involvement of the pelvic sidewall lymph nodes (PSW) can optionally be considered.
* ECOG status ≤ 1
* Being willing and able to give full written consent for participation

Exclusion Criteria:

* Previous rectal cancer treatment
* Previous irradiation to the treatment area e.g. prostate cancer
* Hip prosthesis
* Contraindications to MRI
* Pregnancy
* Abnormal DPYD genotype
* Known contraindication to 5-FU, Capecitabine or Oxaliplatin as judged by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute gastro-intestinal toxicity equal or higher than grade 2 | Up to administration of the last course of chemotherapy or week 22, whichever comes first
  Incidence of acute gastro-intestinal toxicity from therapy graded according to CTCAE ver. 5.

SECONDARY OUTCOMES:
Number of participants that require alteration of chemotherapy due to toxicity | From treatment week 3 up to week 20
  Alterations of chemotherapy, defined as dose-reduction or pre-maturely stopping chemotherapy administration
Number of patients with disease related treatment failure | 5 years after surgery
  Disease-related treatment failure include the first of any of the following events:
  (i) During treatment: Non-radical resection of primary tumor (R2 resection) or un-fit of for surgery due to progression, death from treatment (ii) During, or after treatment: Loco-regional recurrence (including regrowth after potential watch-and-wait), distant metastasis (including M re-staging at surgery), death from rectal cancer, second primary rectal cancer.
Number of patients with pathological complete response (pCR) | At surgery i.e. in treatment week 23-28
  pCR after completion of the intended or tolerated TNT
Tumour regression grade | Baseline to response evaluation on MR in up to week 25 of the study
  Radiological based clinical response evaluation on MR (mrTRG)
Overall survival | Follow-up until 5 years or death
  Overall survival from time of inclusion until death
Incidence of late gastro-intestinal toxicity equal or higher than grade 2 | 5 years
  Incidence of late gastro-intestinal events (e.g.diarrhea, rectal hemorrhage, rectal and/or abdominal pain) from therapy graded according to CTCAE ver. 5.

OTHER OUTCOMES:
Bowel exposure | Treatment week 1-2
  Radiation dose to bowel
Immunogenic alterations from TNT | Baseline and at surgery i.e. in treatment week 23-28
  Presence of selected immune cells
Perfusion changes on MR | Baseline and at MR response evaluation up to week 25 of the study
  Changes in perfusion from contrast-enhanced MR
Diffusion changes on MR | Baseline and at MR response evaluation up to week 25 of the study
  Changes in diffusion from diffusion-weighted MR
Patient reported general outcome measures | Baseline and up to 5 years of the study
  Quality of life using EORTC qlq-c30 questionnaire
Patient reported colo-rectal outcome measures | Baseline and up to 5 years of the study
  Quality of life using EORTC qlq-cr29 questionnaire
Patient reported bowel-related outcome measures | Baseline and up to 5 years of the study
  Quality of life using low anterior resection syndrome (LARS) score

CONTACTS AND LOCATIONS:
Overall Officials: Unn Hege Lilleøren, MD, Principal Investigator — Dept. of Oncology and Medical Physics, Haukeland University Hospital, Bergen, Norway
Locations (1):
- Haukeland University Hospital, Bergen, Norway